CLINICAL TRIAL: NCT04158076
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase III Trial to Evaluate the Efficacy and Safety of Co-administrated AD-2071 and AD-2073 in Patients With Primary Hypercholesterolemia and Essential Hypertension
Brief Title: Evaluating the Efficacy and Safety of Co-administrated Rosuvastatin/Ezetimibe and Telmisartan/Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROZETELA RCT
Record Dates: First submitted 2019-11-07; First posted 2019-11-08 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Hypercholesterolemia; Hypertension | interventions — Ezetimibe; Rosuvastatin Calcium; Telmisartan; Amlodipine; telmisartan amlodipine combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-administered of AD-2071 and AD-2073 (Experimental): 48 subjects will be assigned and the subjects will be administered "AD-2071(Ezetimibe/Rosuvastatin) and AD-2073(Telmisartan/Amlodipine)" for 8 weeks.
  Interventions: Drug: Ezetimibe/Rosuvastatin; Drug: Telmisartan/Amlodipine 80 Mg-5 Mg ORAL TABLET
- Co-administered of AD-2071 and AD-2072 (Active Comparator): 48 subjects will be assigned and the subjects will be administered "AD-2071(Ezetimibe/Rosuvastatin) and AD-2072(Telmisartan)" for 8 weeks.
  Interventions: Drug: Ezetimibe/Rosuvastatin; Drug: Telmisartan
- AD-2073 (Active Comparator): 48 subjects will be assigned and the subjects will be administered "AD-2073(Telmisartan/Amlodipine)" for 8 weeks.
  Interventions: Drug: Telmisartan/Amlodipine 80 Mg-5 Mg ORAL TABLET

INTERVENTIONS:
Drug: Ezetimibe/Rosuvastatin — PO, Once daily(QD), 8weeks
  Other Names: Rosuvamibe Tab.
  Arms: Co-administered of AD-2071 and AD-2072; Co-administered of AD-2071 and AD-2073
Drug: Telmisartan — PO, Once daily(QD), 8weeks
  Other Names: Micardis Tab.
  Arms: Co-administered of AD-2071 and AD-2072
Drug: Telmisartan/Amlodipine 80 Mg-5 Mg ORAL TABLET — PO, Once daily(QD), 8weeks
  Other Names: Twynsta
  Arms: AD-2073; Co-administered of AD-2071 and AD-2073

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of co-administrated Rosuvastatin/Ezetimibe and Telmisartan/Amlodipine in patients with primary hypercholesterolemia and essential hypertension.

DETAILED DESCRIPTION:
This trial is a phase 3 study to evaluate efficacy and safety of co-administrated Rosuvastatin/Ezetimibe and Telmisartan/Amlodipine in patients with primary hypercholesterolemia and essential hypertension.

In "Rosuvastatin/Ezetimibe+Telmisartan/Amlodipine" treatment group, 48 subjects will be assigned and the subjects administer "Rosuvastatin/Ezetimibe+Telmisartan/Amlodipine" for 8 weeks.

In "Rosuvastatin/Ezetimibe +Telmisartan " treatment group, 48 subjects will be assigned and the subjects administer "Rosuvastatin/Ezetimibe+Telmisartan" for 8 weeks.

In "Telmisartan/Amlodipine" treatment group, 48 subjects will be assigned and the subjects administer "Telmisartan/Amlodipine" for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects with hypertension and hyperlipidemia

Exclusion Criteria:

* Patient with known or suspected secondary hypertension
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Low density lipoprotein cholesterol (LDL-C) | Baseline, Week 8
  LDL-C change at Week 8 compared AD-2071 + AD-2073 with AD-2073
Mean sitting systolic blood pressure (MSSBP) | Baseline, Week 8
  MSSBP change at Week 8 compared AD-2071 + AD-2072 with AD-2071 + AD-2073

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Soo Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No